CLINICAL TRIAL: NCT00088647
Title: A Phase 1 Dose-Escalation Study of Intravenous MST-997 Formulated in Intralipid 20% Administered Weekly in Subjects With Advanced Malignant Solid Tumors
Brief Title: Study Evaluating MST-997 in Advanced Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 3161K1-100
Record Dates: First submitted 2004-07-30; First posted 2004-08-02 (Estimated); Last update posted 2006-12-08 (Estimated); Status verified 2006-12

CONDITIONS: Neoplasms
Keywords: advanced malignant solid tumors; breast cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — MST 997

INTERVENTIONS:
Drug: MST-997

SUMMARY:
The primary objective of this clinical research study is to evaluate the safety, tolerability, and maximum tolerated dose (MTD) of intravenous (IV) MST-997 formulated in Intralipid 20% administered on a weekly schedule to subjects with advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Documented histological or cytological diagnosis confirming the presence of malignant solid tumor
* Tumor progression after conventional therapy for cancer or a malignant solid tumor for which no conventional therapy exists
* Subjects enrolled in the MTD confirmation cohort should have a documented histologic and/or cytologic diagnosis of metastatic breast cancer or non-small cell lung cancer (NSCLC) and should not have received more than 2 prior chemotherapy regimens for metastatic disease (adjuvant and neoadjuvant chemotherapy will not be included in the maximum of 2 prior regimens described above)

Exclusion Criteria:

* Subjects with symptomatic or clinically active central nervous system (CNS) metastases. Subjects who have had prior treatment with radiotherapy or surgical resection for CNS metastases will be permitted if CNS metastases have remained stable and have not required any treatment for at least 3 months prior to first dose of test article
* History of any other primary malignancy with less than 5 years documentation of a disease-free state (Subjects with a history of basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ, which have been successfully treated, are not excluded)
* Recent major surgery (within 14 days before the first dose) or chemotherapy within 28 days before the first dose of MST-997 (42 days if the previous chemotherapy included nitrosoureas or mitomycin C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
To evaluate the safety, tolerability and MTD of IV MST-997 throughout patients participation on trial.

SECONDARY OUTCOMES:
To obtain preliminary information on the pharmacokinetics (during cycle 1) and antitumor activity of MST-997 (approximately every 8 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (3):
- United States (3):
  - New York, New York
  - Cleveland, Ohio
  - Nashville, Tennessee